CLINICAL TRIAL: NCT04325282
Title: Impact of Repetitive Transcranial Magnetic Stimulation (TMS) on Spike Frequency and Brain Connectivity in Children With Benign Epilepsy With Centrotemporal Spike (BECTS)
Brief Title: Transcranial Magnetic Stimulation for BECTS
Acronym: TMS4BECTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Fiona Baumer, Instructor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 37514; K23NS116110 (NIH)
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Benign Epilepsy With Centrotemporal Spikes; Language Problems; Learning Disorders
Keywords: Transcranial Magnetic Stimulation (TMS); Electroencephalogram (EEG); Children; Pediatric; Interictal Epileptiform Discharges; Brain connectivity
MeSH Terms: conditions — Epilepsy, Rolandic; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Children will receive active repetitive TMS (rTMS) on one day and sham stimulation on a second day. The order of stimulation will be randomized on a per-participant basis.
  Children and parents/guardians will not be told if they are receiving sham or inhibitory rTMS on a given day. The research team will know at the time of stimulation, however, as they will have to choose which coil to use. The TMS-EEG files will be coded and the team member analyzing the files for change in IED (spike) frequency and change in connectivity will be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Children with BECTS (Experimental): Children will receive sham and active rTMS on 2 separate study visits separated by at least 1 week.
  Interventions: Device: Active rTMS; Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — 1Hz rTMS delivered for 15-20 minutes
Device: Sham rTMS — sham rTMS delivered for 15-20 minutes

SUMMARY:
Benign epilepsy with centrotemporal spikes (BECTS) is the most common pediatric epilepsy syndrome. Affected children typically have a mild seizure disorder, but yet have moderate difficulties with language, learning and attention that impact quality of life more than the seizures. Separate from the seizures, these children have very frequent abnormal activity in their brain known as interictal epileptiform discharges (IEDs, or spikes), which physicians currently do not treat. These IEDs arise near the motor cortex, a region in the brain that controls movement.

In this study, the investigators will use a form of non-invasive brain stimulation called transcranial magnetic stimulation (TMS) to determine the impact of IEDs on brain regions important for language to investigate: (1) if treatment of IEDs could improve language; and (2) if brain stimulation may be a treatment option for children with epilepsy.

Participating children will wear electroencephalogram (EEG) caps to measure brain activity. The investigators will use TMS to stimulate the brain region where the IEDs originate to measure how this region is connected to other brain regions. Children will then receive a special form of TMS called repetitive TMS (rTMS) that briefly reduces brain excitability. The study will measure if IEDs decrease and if brain connectivity changes after rTMS is applied.

The investigators hypothesize that the IEDs cause language problems by increasing connectivity between the motor cortex and language regions. The investigators further hypothesize that rTMS will reduce the frequency of IEDs and also reduce connectivity between the motor and language region

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Benign Epilepsy with Centrotemporal Spikes (BECTS), sometimes called Rolandic Epilepsy. Diagnosis will be based on a history of a focal motor seizure (affecting the face or causing hypersalivation) or a history of a seizure out of sleep AND an EEG with unilateral or bilateral centrotemporal spike waves.
* English-speaking

Exclusion Criteria:

* History of prematurity < 35 weeks gestational age;
* History of serious neurologic problems (i.e. history of other seizure disorder other than simple febrile seizure, head trauma with prolonged loss of consciousness, cerebrovascular accident or neuro-inflammatory disease)
* Focal deficits on neurologic exam
* History of abnormal MRI (with clear gray or white matter abnormality)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Baumer, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan.

REFERENCES:
- [Background] Baumer FM, Pfeifer K, Fogarty A, Pena-Solorzano D, Rolle CE, Wallace JL, Rotenberg A, Fisher RS. Cortical Excitability, Synaptic Plasticity, and Cognition in Benign Epilepsy With Centrotemporal Spikes: A Pilot TMS-EMG-EEG Study. J Clin Neurophysiol. 2020 Mar;37(2):170-180. doi: 10.1097/WNP.0000000000000662. PMID 32142025
- [Background] Mishra A, Maiti R, Mishra BR, Jena M, Srinivasan A. Effect of Repetitive Transcranial Magnetic Stimulation on Seizure Frequency and Epileptiform Discharges in Drug-Resistant Epilepsy: A Meta-Analysis. J Clin Neurol. 2020 Jan;16(1):9-18. doi: 10.3988/jcn.2020.16.1.9. PMID 31942753
- [Background] Chen R, Spencer DC, Weston J, Nolan SJ. Transcranial magnetic stimulation for the treatment of epilepsy. Cochrane Database Syst Rev. 2016 Aug 11;(8):CD011025. doi: 10.1002/14651858.CD011025.pub2. PMID 27513825
- [Result] She X, Qi W, Nix KC, Menchaca M, Cline CC, Wu W, He Z, Baumer FM. Repetitive transcranial magnetic stimulation modulates brain connectivity in children with self-limited epilepsy with centrotemporal spikes. Brain Stimul. 2025 Mar-Apr;18(2):287-297. doi: 10.1016/j.brs.2025.02.018. Epub 2025 Feb 24. PMID 40010636
- [Result] She X, Nix KC, Cline CC, Qi W, Tugin S, He Z, Baumer FM. Stability of transcranial magnetic stimulation electroencephalogram evoked potentials in pediatric epilepsy. Sci Rep. 2024 Apr 20;14(1):9045. doi: 10.1038/s41598-024-59468-8. PMID 38641629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with Self Limited Epilepsy with Centrotemporal Spikes (SeLECTS), formerly known as Benign Epilepsy with Centrotemporal Spikes (BECTS).
Groups:
- Children With SeLECTS - Active, Then Sham rTMS; Children With SeLECTS - Sham, Then Active rTMS: Children will receive sham and active (1 Hz) rTMS on 2 separate study visits separated by at least 1 week.
Period: First Intervention (1 Day)
Arm/Group | Children With SeLECTS - Active, Then Sham rTMS | Children With SeLECTS - Sham, Then Active rTMS
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period (1 Week)
Arm/Group | Children With SeLECTS - Active, Then Sham rTMS | Children With SeLECTS - Sham, Then Active rTMS
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Children With SeLECTS - Active, Then Sham rTMS | Children With SeLECTS - Sham, Then Active rTMS
Started | 11 | 10
Completed | 11 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants with Analyzable Data (Remained awake for both active & sham rTMS sessions)
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With SeLECTS - Active, Then Sham rTMS | Children With SeLECTS - Sham, Then Active rTMS | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (1.4) | 10.1 (1.8) | 9.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 4 | 14
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Interictal Epileptiform Discharge (IED) Frequency
Description: We will count the number of IEDs/minute before and after application of active rTMS as well as before and after sham rTMS. We will compare the change in IEDs induced by the active and sham stimulation.
Time Frame: Before and after intervention (approximately 4 hours/visit on 2 study days one week apart)
Population: Participants with Analyzable Data (Remained awake for both active & sham rTMS sessions)
Measure: Median (Inter-Quartile Range); unit: IEDs per 5 minutes
Groups:
- Children With SeLECTS - Active rTMS; Children With SeLECTS - Sham rTMS: Children will receive sham and active (1 Hz) rTMS on 2 separate study visits separated by at least 1 week.
Arm/Group | Children With SeLECTS - Active rTMS | Children With SeLECTS - Sham rTMS
Number analyzed (Participants) | 19 | 19
IEDs per 5 minutes
  Before rTMS | 0 [0 to 20.5] | 0 [0 to 18]
  After rTMS | 0 [0 to 12] | 0 [0 to 18.5]
  Change from pre-rTMS to post-rTMS | 0 [-6.5 to 0] | 0 [-1 to 0]
Statistical Analysis 1: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change after active rTMS (post-rTMS compared to pre-rTMS); Test type: Other; p = 0.04, Wilcoxon signed rank test — The a priori threshold for statistical significance was <0.05
Statistical Analysis 2: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change after sham rTMS (post-rTMS compared to pre-rTMS); Test type: Other; p = 0.46, Wilcoxon signed rank test — The a priori threshold for statistical significance was <0.05
Statistical Analysis 3: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change induced by active rTMS versus sham rTMS; Test type: Other; p = 0.12, Wilcoxon signed rank test — The a priori threshold for statistical significance was <0.05

2. Secondary Outcome: Change in Brain Connectivity
Description: We will measure brain connectivity before and after application of active rTMS as well as before and after sham rTMS. We will compare the change in connectivity induced by the active and sham stimulation. In particular, we will look at how connectivity changes between the motor cortex and language regions of the brain. We chose 3 regions of interest per hemisphere (-F: Frontal, -M: Motor, -T: Temporal). rTMS was applied to the hemisphere with more spikes on clinical EEG, and hence all regions were further qualified as being ipsilateral (i-) or contralateral (c-) to rTMS application.
  Connectivity is measured in the weighted Phase Lag Index (wPLI) in the beta-frequency band, a phase-based connectivity measure which runs from a theoretical minimum of 0 (no connectivity) to 1 (complete connectivity).
Time Frame: Before and after intervention (approximately 4 hours/visit on 2 study days one week apart)
Population: Participants with Analyzable Data (Remained awake for both active & sham rTMS sessions)
Measure: Median (Inter-Quartile Range); unit: wPLI
Arm/Group | Children With SeLECTS - Active rTMS | Children With SeLECTS - Sham rTMS
Number analyzed (Participants) | 19 | 19
wPLI
  Change in cF-iT Connectivity | -0.025147033 [-0.06736053235 to -0.009095556347] | 0.001240549 [-0.01674470333 to 0.03546101011]
  Change in cM-iT Connectivity | -0.026464821 [-0.09033280758 to -0.004439810119] | 0.015413055 [-0.009845339466 to 0.05680533952]
  Change in iF-cM Connectivity | -0.038566551 [-0.07507071808 to -0.000831546384] | 0.009032342 [-0.01706492182 to 0.02160196731]
  Change in iF-iT Connectivity | -0.031871907 [-0.06020716415 to -0.008456458479] | 0.005724761 [-0.01917787091 to 0.03179566288]
  Change in iF-cF Connectivity | -0.017828074 [-0.131733617 to -0.005389702698] | 0.004773205 [-0.01693847284 to 0.04093271291]
  Change in iM-cT Connectivity | -0.016437136 [-0.05883184645 to 0.009583756] | 0.010533673 [-0.01520736144 to 0.02572202471]
  Change in iF-cT Connectivity | -0.017946561 [-0.05996626405 to 0.001548810394] | 0.008023921 [-0.005516234384 to 0.02195947435]
  Change in iF-iM Connectivity | -0.028419447 [-0.06790541051 to -0.01930392446] | 0.011937066 [-0.01998846337 to 0.03538472482]
  Change in iT-cT Connectivity | -0.041984947 [-0.08226344292 to 0.00820188987] | -0.000655525 [-0.009649517287 to 0.0352091797]
  Change in cF-cT Connectivity | -0.022140561 [-0.04754855866 to 0.006893751688] | 0.006909577 [-0.01526276726 to 0.03540581226]
  Change in cF-cM Connectivity | -0.011221254 [-0.0543134682 to 0.006043824425] | 0.009773165 [-0.009669095958 to 0.03596951991]
  Change in cF-iM Connectivity | -0.031668097 [-0.05419498148 to 0.003974133567] | 0.01966644 [-0.009877540375 to 0.0318713625]
  Change in iM-iT Connectivity | -0.030898043 [-0.05097858412 to -0.003586219461] | 0.002850137 [-0.004130106912 to 0.02728766311]
  Change in cM-cT Connectivity | -0.029060306 [-0.05558707448 to 0.01102180261] | -0.00727134 [-0.0244931598 to 0.02049569394]
  Change in iM-cM Connectivity | -0.032771045 [-0.07116425937 to 0.004104307197] | 0.004707047 [-0.02741234695 to 0.02510245297]
Statistical Analysis 1: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in cF-iT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — Given the multiple ROIs investigated, we adjusted significance thresholds using principal component analysis, which accounts for the effective number of independent tests. This method is suitable when data in each comparison are not completely independent, as is the case with EEG where signal represents summated activity from multiple regions; p < 0.0001, Wilcoxon signed-rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 2: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in cF-iT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.69, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 3: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in cF-iT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 4: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in cM-iT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 5: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in cM-iT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.43, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 6: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in cM-iT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 7: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iF-cM connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.002, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 8: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iF-cM connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.54, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 9: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iF-cM connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.007, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 10: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iF-iT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.002, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 11: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iF-iT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.32, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 12: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iF-iT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.01, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 13: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iF-cF connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.003, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 14: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iF-cF connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.29, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 15: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iF-cF connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.02, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 16: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iM-cT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.003, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 17: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iM-cT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.66, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 18: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iM-cT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.008, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 19: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iF-cT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.005, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 20: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iF-cT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.87, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 21: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iF-cT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.11, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 22: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iF-iM connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.012, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 23: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iF-iM connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.46, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 24: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iF-iM connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.02, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 25: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iT-cT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.01, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 26: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iT-cT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.99, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 27: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iT-cT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.04, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 28: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in cF-cT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.01, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 29: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in cF-cT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.31, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 30: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in cF-cT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.05, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 31: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in cF-cM connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.03, Wilcoxon signed rank test; The threshold for statistical significance was p < 0.0076
Statistical Analysis 32: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in cF-cM connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.20, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 33: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in cF-cM connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.04, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 34: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in cF-iM connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.05, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 35: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in cF-iM connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.59, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 36: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in cF-iM connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.12, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 37: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iM-iT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.10, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 38: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iM-iT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.57, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 39: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iM-iT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.06, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 40: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in cM-cT connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.12, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 41: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in cM-cT connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.69, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 42: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in cM-cT connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.14, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071
Statistical Analysis 43: Comparison: Children With SeLECTS - Active rTMS; Within-group analysis of change in iM-cM connectivity during active rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.12, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 44: Comparison: Children With SeLECTS - Sham rTMS; Within-group analysis of change in iM-cM connectivity during sham rTMS (post-rTMS versus pre-rTMS); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.60, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0076
Statistical Analysis 45: Comparison: Children With SeLECTS - Active rTMS vs Children With SeLECTS - Sham rTMS; Between-group analysis of change in iM-cM connectivity induced by active versus sham rTMS; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.04, Wilcoxon signed rank test — The threshold for statistical significance was p < 0.0071

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Children With SeLECTS - Active rTMS | Children With SeLECTS - Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 2/19 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Children With SeLECTS - Active rTMS (N=19) | Children With SeLECTS - Sham rTMS (N=19)
Head pain during stimulation (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT04325282/Prot_001.pdf
  • Statistical Analysis Plan (2025-07-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT04325282/SAP_002.pdf
  • Informed Consent Form (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT04325282/ICF_000.pdf